CLINICAL TRIAL: NCT04429035
Title: Inhibition of Aortic Valve Calcification Through the Carboxylation Mechanism of Matrix Gla Protein (MGP), Following Administration of Vitamin K2 (Menaquinone-7). Correlation With Mitral Annulus and Ascending Aorta Calcification.
Brief Title: SLOW-Slower Progress of caLcificatiOn With Vitamin K2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Konstantinos Toutouzas, Professor of Cardiology, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 55461
Record Dates: First submitted 2020-05-31; First posted 2020-06-11 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Calcification; Mitral Annular Calcification; Mitral Valve Calcification; Mitral Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve, Calcification of; Mitral Valve Stenosis | interventions — Vitamin K 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin K2 (Experimental): Participants receive Vitamin K2 (Menaquinone) 100mcg tablet orally 3 times daily for 12 months.
  Interventions: Dietary Supplement: Vitamin K2
- Placebo (Placebo Comparator): Participants receive Vitamin K2 (Menaquinone) placebo tablet matching Vitamin K2 (Menaquinone) orally 3 times daily for 12 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin K2 — Administration of 300 μg Vitamin K2 (MQ7) daily p.o
  Arms: Vitamin K2
Dietary Supplement: Placebo — Administration of 300 μg Vitamin K2 (MQ7) Placebo daily p.o
  Arms: Placebo

SUMMARY:
A randomized 12-month trial will include two groups of 100 individuals aged over 50 years, with asymptomatic mild to moderate Aortic valve stenosis (AVA > 1 cm2, Vmax < 4 m/s). The first group of 100 individuals will serve as the intervention group that will receive 300 mcg of K2 vitamin on a daily basis, while the second group of 100 individuals will be the control group that will receive placebo on a daily basis as well. Both groups will be monitored identically in order to investigate therapeutic effects on calcification and valve stenosis progression. Correlation with Mitral annulus and ascending Aorta.Exclusion criteria: Chronic Kidney disease, Vitamin K antagonists, statins, age < 50 y.o,prosthetic valves,Aortic Valve area (AVA) < 1cm2 ,Vmax > 4 m/s

DETAILED DESCRIPTION:
For the purposes of this study, all individuals will be subjected to the same quantitative and qualitative tests, before and after the daily administration of 300mcg K2 vitamin/placebo for a period of one year.Clinical examination,extensive blood laboratory tests,direct measurement of Dephosphorylated-uncarboxylated MGP(dp-ucMGP), Echocardiogram and ECS,carotid ultrasound,ophthalmologic exam,further imaging methods with MSCT Calcium Score(Agatston score) will take place.Correlations with their medical and pharmacological therapy history.

Before and after the administration of VK2/placebo, the following measurements will take place i)Quantitative and percentile rate determination of Aortic Valve, Mitral Valve and Ascending Aorta calcification via MSCT Calcium score without contrast.

ii)Echocardiogram and calcification evaluation via Echocardiographic Calcium Score (ECS), iii)Determination of changes in carotid intima-media thickness (cIMT) and Carotid stenosis iv)Standard ophthalmologic examination v)Direct measurement of Dephosphorylated-uncarboxylated MGP(dp-ucMGP) vi)Correlation with blood biomarkers

ELIGIBILITY:
Inclusion Criteria:

* ASYMPTOMATIC AV STENOSIS WITH AVA>1 cm2 & Vmax<4m/s

Exclusion Criteria:

* AVK,STATINS,MSCT THE LAST 6 MONTHS,PROSTHETIC VALVES, AVA<1 cm2,Vmax>4m/s

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-09-23 (Actual); Primary Completion 2022-10-23 (Estimated); Study Completion 2023-12-23 (Estimated)

PRIMARY OUTCOMES:
Evaluation of calcification change of Aortic valve.Correlation With Mitral annulus and ascending Aorta calcification.A randomized 12-month trial. | Each patient will be evaluated twice a year.Once before the administartion of VK2/Placebo and after a period of a 12 month administration of VK2/PLACEBO
  The calcification change will be evaluated via a 64 MSCT scanner measuring the calcium via Agatston score, before and after administration of VK2/placebo.The following measurements will take place and after 12 months will be compared.

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - First Department of Cardiology, University of Athens, Athens, Attica
  - Hippokration Hospital 1st Department of Cardiology,National and Kapodistrian University of Athens,Medical School, Athens, Attica